CLINICAL TRIAL: NCT07404969
Title: An Interventional Study Evaluating Telomere and Biological Aging Hallmarks Profiling to Guide an Integrative Traditional Chinese and Conventional Medicine Approach in Women With Post-Treatment Unexplained Infertility
Brief Title: Biological Aging Hallmarks-Guided Integrative TCM and Conventional Medicine in Post-Treatment Unexplained Female Infertility
Acronym: TECMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BEYOND GENOMiX SA, AG, Ltd (Industry)
Collaborators: Praxis für Akupunktur und Chinesische Arzneimittel (Unknown); Fertisuisse Ltd, SA, AG (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGX-INFERT-TEL-TCM-2025; 70596.1 INNO-LS (Other Grant/Funding Number: Innosuisse)
Record Dates: First submitted 2025-12-18; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Idiopathic Infertility; Infertility Unexplained; Infertility (IVF Patients); Infertility Assisted Reproductive Technology; Infertility Female
Keywords: Telomere dysfunction; Telomere attrition; Telomere biology; Cellular aging; Mitochondrial dysfunction; Cellular senescence; Reproductive aging; Functional infertility; Idiopathic infertility; Post-treatment unexplained infertility; Oocyte quality; Endometrial receptivity; Biomarkers of reproductive quality; Single-cell FISH; Leukocyte telomere length; Molecular etiology of infertility; Aging hallmarks; Traditional Chinese Medicine; Integrative fertility therapy; Nutraceutical support; Mitochondrial biogenesis; Oxidative stress; Reproductive resilience; Beyond Genomix
MeSH Terms: conditions — Infertility; Infertility, Female; Mitochondrial Diseases | interventions — Reproductive Techniques, Assisted

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open-label interventional study evaluating a personalized telomere-guided therapeutic approach in women with post-treatment unexplained (functionally idiopathic) infertility. Each participant receives an individualized integrative protocol tailored to her telomere molecular profile and interconnected aging hallmarks, including mitochondrial dysfunction and cellular senescence.
  The intervention combines TCM formulations with targeted nutraceutical support to restore telomere integrity, enhance mitochondrial activity, and reduce senescence, as reflected by the percentage of super-short telomeres (<5 kb). The study includes three phases: baseline telomere and reproductive assessment, a 4-12 week preconception phase with personalized therapy, and a conception phase (natural or ART) under continued integrative care.
  The primary outcome is the restoration of reproductive quality through telomere and related pathways rejuvenation, to improve oocyte competence.
Masking Description: This is an open-label study. No parties are masked to the intervention. Participants, investigators, and assessors are aware of the assigned treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological Aging-Informed Integrative Fertility Intervention (Experimental): Participants assigned to this arm undergo a baseline reproductive evaluation and molecular profiling related to biological aging, including leukocyte telomere analysis. Women presenting biological aging-related molecular signatures complete a personalized preconception integrative intervention lasting 4 to 12 weeks prior to natural conception attempts or IUI / IVF.
  The intervention combines individualized botanical formulations derived from TCM and targeted nutraceutical supplementation, administered alongside standard fertility care. These interventions are intended to support telomere-related cellular integrity, mitochondrial function, regulation of cellular senescence associated pathways, oxidative balance, and overall tissue homeostasis.
  Following the preconception phase, participants proceed with natural conception attempts or ART while continuing the integrative support. Clinical pregnancy outcomes & changes in molecular and reproductive parameters are prospectively assessed.
  Interventions: Other: 1. Aging Hallmarks Biomarker Profiling (Telomere-Based); Other: 2. Integrative Botanical and Nutraceutical Intervention; Procedure: 3. Natural Conception or Assisted Reproductive Technologies

INTERVENTIONS:
Other: 1. Aging Hallmarks Biomarker Profiling (Telomere-Based) — Participants undergo baseline molecular profiling of biological aging biomarkers derived from the hallmarks of aging framework, with a primary focus on telomere-related parameters measured in peripheral blood leukocytes. Telomere analysis includes assessment of mean telomere length, the percentage of critically short ("super-short") telomeres, and telomere-length distribution profiles.
  Together, these biomarkers provide a measure of biological age and define molecular signatures of cellular aging relevant to ovarian and reproductive tissue function, including processes associated with telomere attrition, cellular senescence, and downstream aging hallmarks. Molecular parameters are assessed at baseline and, where applicable, longitudinally according to the study protocol for stratification and monitoring purposes.
Other: 2. Integrative Botanical and Nutraceutical Intervention — Participants receive a personalized integrative intervention consisting of botanical formulations derived from Traditional Chinese Medicine (TCM) and targeted nutraceutical supplementation during a preconception period of 4 to 12 weeks. The intervention is administered alongside standard fertility care and is informed by biological aging-related molecular signatures. The integrative support is intended to address biological processes associated with aging hallmarks, including telomere-related cellular integrity, mitochondrial function, cellular senescence-associated pathways, oxidative balance, and tissue homeostasis.
Procedure: 3. Natural Conception or Assisted Reproductive Technologies — Following completion of the preconception phase and confirmation of stabilization of biological aging-related molecular profiles associated with the hallmarks of aging, participants proceed to conception attempts either through natural cycles or through assisted reproductive technologies, including intrauterine insemination (IUI) or in vitro fertilization (IVF), according to clinical indication. Assisted reproductive procedures are conducted in accordance with standard clinical practice and local guidelines. The choice of conception method is determined by routine clinical criteria and participant preference. No experimental modifications to standard ART protocols are introduced as part of this intervention.

SUMMARY:
The goal of this clinical trial is to determine whether telomere profiling and other biological aging hallmarks can help identify underlying mechanisms of persistent infertility in women with post-treatment unexplained infertility. The study also evaluates whether a personalized integrative treatment guided by these biomarkers can improve reproductive outcomes.

The study includes women aged 25 to 42 years who continue to experience infertility despite appropriate management of identifiable reproductive conditions and repeated attempts with assisted reproductive technologies (ART), such as intrauterine insemination (IUI) or in vitro fertilization (IVF).

The main questions this study aims to answer are:

* Can telomere and biological aging hallmarks profiling identify a biological aging phenotype associated with infertility?
* Can an integrative treatment guided by these profiles improve clinical pregnancy outcomes?

Participants will:

* Undergo a baseline reproductive evaluation and blood-based assessment of telomeres and aging hallmarks.
* Receive an integrative approach combining Traditional Chinese Medicine (TCM), targeted nutritional support, and standard fertility care.
* Proceed with natural conception attempts or standard assisted reproductive technologies following the preconception phase.
* Participants will be followed to assess pregnancy outcomes and changes in biological aging hallmarks.

DETAILED DESCRIPTION:
1. Scientific Background and Clinical Need

   Infertility affects approximately one in six couples worldwide. In up to 40 percent of cases, no clear etiology can be identified even after comprehensive clinical and laboratory evaluation, a condition traditionally defined as idiopathic infertility. In parallel, a growing number of women experience persistent reproductive failure despite adequate management of identifiable conditions such as endometriosis, polycystic ovary syndrome, or hormonal imbalance. This category, referred to as post-treatment unexplained or functionally idiopathic infertility, includes patients whose anatomical and endocrine parameters appear normalized, yet who continue to experience repeated ART failures, whether through intrauterine insemination or in vitro fertilization.

   Both idiopathic and post-treatment unexplained infertility reveal a fundamental limitation of current diagnostic frameworks. Conventional assessments may normalize structural or hormonal parameters while overlooking deeper molecular dysfunctions that impair reproductive capacity.

   Emerging evidence suggests that many of these cases correspond to an unrecognized form of reproductive aging, in which cellular and molecular decline within reproductive tissues occurs earlier than chronological aging would predict. In other words, the reproductive system becomes biologically older than the patient's calendar age.

   Conventional diagnostic tools primarily assess quantitative and structural parameters such as hormonal levels, oocyte count, uterine morphology, or tubal patency. However, these metrics fail to capture the qualitative dimensions of cellular health, particularly those associated with the hallmarks of aging such as telomere erosion, mitochondrial dysfunction, and cellular senescence.

   This diagnostic gap underscores the need for molecular biomarkers capable of reclassifying idiopathic infertility into a biologically defined and actionable condition, enabling both mechanistic understanding and targeted therapeutic intervention.
2. The Hallmarks of Aging and the Central Role of Telomeres

   Aging is now understood through the framework of biological hallmarks, a unified model describing the processes that collectively drive functional decline. These hallmarks are categorized into primary, secondary, and tertiary groups:

   2.1. Primary hallmarks: the initiating sources of molecular damage, including genomic instability, telomere attrition, epigenetic alterations, and loss of proteostasis.

   2.2. Secondary hallmarks: the cellular responses to this damage, such as mitochondrial dysfunction, cellular senescence, and deregulated nutrient sensing.

   2.3. Tertiary hallmarks: the downstream manifestations of chronic cellular stress, including altered intercellular communication and chronic inflammation.

   This hierarchy functions as a domino-like system, in which the perturbation of the primary hallmarks initiates secondary and tertiary responses that progressively erode tissue homeostasis and ultimately lead to age-related disease. When this process unfolds in the brain, it manifests as neurodegeneration; when it occurs in the ovaries, it accelerates reproductive aging and loss of fertility.

   At the base of this biological network lies telomere biology, which serves as both a sensor and structural foundation of cellular aging. Among all primary hallmarks, telomere attrition occupies a pivotal and initiating position, as it represents the most direct and quantifiable indicator of cumulative molecular stress. Its destabilization propagates dysfunction across multiple downstream hallmarks, activating mitochondrial decline, genomic instability, cellular senescence, and chronic inflammation. In this sense, telomere erosion forms the base of the aging cascade, upon which secondary and tertiary hallmarks unfold, eventually leading to age-related diseases when the process remains uncorrected.
3. Telomere

   Imagine the genome as a book, with telomeres serving as its protective covers, keeping the pages intact and preventing them from fraying. With each cell division, these covers naturally wear down in somatic cells, where telomerase activity is limited to absent, making gradual telomere shortening an intrinsic feature of cellular aging. In contrast, germline cells and certain stem cell populations express telomerase and other maintenance mechanisms that help preserve telomere length, ensuring genomic stability across generations.

   However, when oxidative stress or replicative demand exceeds repair capacity, telomere erosion accelerates even in these lineages, compromising chromosomal integrity. As telomeres, the book covers, shorten, the remaining DNA, including the coding genome, which represents about one percent of total DNA, becomes increasingly susceptible to strand breaks, instability, and loss. This phenomenon is systemically reflected in leukocytes, where telomere length provides a measurable proxy for biological aging and cumulative molecular stress across tissues.

   This conceptual analogy translates directly into molecular reality. Telomeres are repetitive DNA sequences located at the tips of chromosomes, where they preserve genome integrity by preventing end-to-end fusions and inappropriate DNA repair signaling. When telomeres become critically short, cells lose their ability to divide safely. Under normal circumstances, such cells either activate repair pathways or undergo programmed cell death (apoptosis).

   When these safety mechanisms fail, cells enter senescence, a non-dividing yet metabolically active state. Senescent cells release inflammatory cytokines and reactive oxygen species, gradually creating a microenvironment of chronic inflammation and oxidative stress. One of the earliest and most profound consequences of this state is mitochondrial decline, a process intimately linked to the telomere damage response pathway. Dysfunctional telomeres trigger persistent DNA damage signaling that alters mitochondrial biogenesis and energy metabolism through the p53-PGC-1α axis, leading to reduced ATP production, elevated reactive oxygen species, and further telomere erosion. Over time, this self-reinforcing loop between telomere instability and mitochondrial dysfunction erodes tissue homeostasis, impairs organ performance, and contributes to the progression of age-related diseases. Thus, telomere shortening is not merely a marker of aging, it is a causal driver of biological decline, linking genomic instability, mitochondrial failure, and systemic dysfunction.

   In reproductive medicine, the decline in fertility is not determined solely by the number of gametes but by their quality, which depends on the health of their surrounding microenvironment. In the context of this clinical study, which focuses on women, this principle is illustrated through the biology of the oocyte and its companion somatic cells. One major determinant of oocyte quality is telomere erosion within granulosa cells, which orchestrate follicular maturation and provide the molecular and metabolic support necessary for meiotic progression. These cells synthesize growth factors, cytokines, and mitochondrial substrates essential for chromosomal stability and cytoplasmic competence. When telomeres in granulosa cells become critically short, the resulting telomere damage response disrupts transcriptional regulation and mitochondrial function, reducing the production of proteins and signaling molecules required for oocyte maturation. As a result, the ovarian reserve may appear quantitatively normal, yet fertilization and embryonic development fail due to impaired oocyte quality.

   Recent studies have shown that shortened telomeres or reduced telomerase activity in granulosa cells correlate with poor oocyte maturation, lower fertilization rates, and diminished embryo quality, even among young women with normal hormonal profiles. This suggests that premature telomere attrition represents a hidden molecular etiology of infertility, where accelerated cellular aging within the follicular niche compromises reproductive potential.

   A similar process occurs directly within oocytes, which are exceptionally long-lived germ cells formed during fetal development and maintained in meiotic arrest for decades. This prolonged quiescence makes them uniquely vulnerable to the cumulative effects of oxidative stress and telomere erosion. As telomeres in oocytes progressively shorten or become structurally unstable, checkpoint pathways are activated, leading to errors in chromosomal segregation, spindle abnormalities, and reduced fertilization potential. Telomere damage also disrupts mitochondrial homeostasis and ATP production, impairing cytoplasmic maturation and early embryonic development. Thus, telomere attrition within oocytes represents a cell-intrinsic mechanism of reproductive aging, complementing the somatic contribution of granulosa cell dysfunction and jointly determining overall oocyte quality.
4. Telomeres as etiology Biomarkers of Reproductive Aging

   Telomeres have been increasingly validated by scientific evidence as qualitative biomarkers of reproductive cellular aging, capturing both the extent and the pattern of molecular decline. Beyond their absolute length, it is the architecture and distribution of telomere lengths across individual cells, and particularly the presence and frequency of critically short telomeres, that define a distinct molecular signature of cellular aging.

   Such signatures cannot be captured through population-averaged measurements, as they only emerge when telomeres are analyzed cell by cell, revealing the intrinsic heterogeneity that determines genomic stability and biological integrity. These distributional profiles serve as early indicators of molecular imbalance: when a subset of cells accumulates ultra-short telomeres, it uncovers the onset of genomic instability and mitochondrial decline long before mean telomere values begin to change.

   Despite this growing understanding, most studies assessing telomere length in infertility have relied on population-averaged techniques such as quantitative PCR (qPCR) or Southern blot. These methods provide only a single mean value across hundreds of cells, masking the subset harboring critically short telomeres, the true initiators of genomic instability, mitochondrial failure, and cellular senescence.

   Moreover, qPCR-based assays suffer from technical variability, including amplification bias, primer inefficiency, and normalization errors, further diluting biological precision. Consequently, the inconsistencies reported in clinical findings reflect not the invalidity of telomere biology, but the limitations of low-resolution technologies incapable of detecting the true pathological pattern.

   To overcome these constraints, this clinical study employs the BEYOND GENOMiX patented single-cell fluorescence in situ hybridization (FISH) protocol, which quantifies telomere length at cellular resolution in leukocytes obtained from peripheral blood. This approach yields both quantitative and qualitative data, mapping the full telomere-length spectrum, exposing cell-to-cell variability, and identifying the subset of cells with critically short telomeres invisible to bulk assays. Results are interpreted individually and benchmarked against age-matched healthy reference ranges.

   The resulting telomere signature is defined by three complementary parameters:

   4.1 Average Telomere Length

   Average telomere length has long been used as a basic metric of cellular aging. It provides an estimate of biological age, but it remains limited: two individuals may display identical mean telomere lengths while exhibiting markedly different cellular and clinical outcomes. This discrepancy arises because average measurements obscure the critical subset of cells harboring extremely short telomeres, those most responsible for genomic instability, mitochondrial dysfunction, cellular senescence, and systemic decline.

   In the context of idiopathic infertility, published studies have reported contradictory results. Some have shown that women with unexplained infertility exhibit significantly shorter mean telomere lengths compared with fertile controls, suggesting premature reproductive aging. Other investigations, however, have found no difference in average telomere length between fertile and infertile cohorts, or even overlapping distributions.

   These inconsistencies likely stem not from biological variability but from the limitations of population-averaged techniques such as qPCR and Southern blot, which cannot distinguish distributional heterogeneity or detect the small proportion of cells carrying critically short telomeres. Consequently, while mean telomere length provides a rough estimate of biological age, it fails to capture the telomere dynamics that determine functional reproductive capacity.

   4.2 Telomere Distribution and Molecular Architecture

   Beyond absolute average length, the distribution and architecture of telomeres across individual cells provide the most biologically meaningful insight into cellular aging. In a healthy state, telomere length follows a balanced distribution, with most cells maintaining intermediate lengths and a minority carrying short or long extremes. This equilibrium reflects effective telomere maintenance, genomic stability, and healthy cellular turnover.

   When the distribution becomes skewed, characterized by a higher fraction of super-short telomeres (defined as shorter than 5 kb), it indicates replicative stress, oxidative injury, or telomerase insufficiency. These critically short telomeres are biologically decisive, as they act as persistent DNA damage signals, activating p53-mediated pathways that suppress mitochondrial regulators PGC-1α/β and disrupt energy metabolism. The result is a cascade of mitochondrial dysfunction, ATP depletion, and reactive oxygen species (ROS) accumulation. Over time, this triggers cellular senescence, stem-cell exhaustion, and chronic inflammation, the systemic consequences of accelerated aging.

   This altered telomere distribution is suggested to represent both a diagnostic signature and a mechanistic driver of reproductive decline, linking nuclear instability with mitochondrial impairment and endocrine dysregulation. Evidence from scientific studies indicates that telomere-length distributions differ between fertile and infertile women, with fertile individuals showing a balanced, Gaussian-like profile dominated by intermediate telomere lengths. In contrast, idiopathically infertile women have been reported to display a left-shifted and compressed distribution, suggesting global telomere shortening. These findings suggest that telomere distribution patterns act as emerging biomarkers of reproductive aging.

   4.3 Critically Short (Super-Short) Telomeres:

   Critically short telomeres, defined as telomere lengths shorter than 5 kb, represent the most decisive point at which genomic stability can no longer be maintained. Such short telomeres lead to mitochondrial dysfunction, ATP depletion, and accumulation of reactive oxygen species (ROS), cellular senescence, stem-cell exhaustion, and chronic inflammation, reflecting the systemic consequences of accelerated aging. The proportion of cells carrying super-short telomeres therefore constitutes a sensitive and quantitative indicator of biological aging. A high fraction of such cells signifies cumulative molecular stress and predicts functional decline at the tissue and organ levels. Evidence shows that it is the presence and proportion of these critically short telomeres, rather than the mean value, that best correlates with genomic instability and functional deterioration. In reproductive biology, this translates into a measurable cellular phenotype that could predict reduced oocyte competence, impaired embryonic development, and diminished implantation potential. Accordingly, this study applies single-cell quantitative analysis to determine the percentage of super-short telomeres in leukocytes, as a proxy for systemic cellular aging.
5. Therapeutic Strategy: Integrative Restoration of Telomere Health

The women enrolled in this study had a documented pattern of treatment resistance, defined by repeated failure of assisted reproductive technologies (ART) and other conventional interventions, despite adequate correction of identified reproductive conditions. Their Telomere profiling performed prior to therapy revealed a molecular signature consistent with those previously described in the literature among idiopathically infertile women, including in studies conducted using the same single-cell FISH platform for telomere analysis as used here. These profiles showed a reduction in mean telomere length, a compressed and left-shifted telomere-length distribution, and a statistically significant enrichment of super-short telomeres (< 5 kb) relative to age matched fertile controls.

On the basis of these molecular findings, participants were selected to test the study's central hypothesis: that restoring telomere integrity, and consequently the downstream cascade of aging hallmarks, could re-establish the biological conditions required for conception.

The study's therapeutic design specifically addressed the three interconnected molecular processes at the core of reproductive aging: telomere erosion, mitochondrial dysfunction, and cellular senescence. These mechanisms form a self-reinforcing cycle in which telomere instability triggers mitochondrial decline through the p53-PGC-1α pathway, leading to reduced biogenesis and elevated oxidative stress, which in turn accelerates telomere shortening and induces premature senescence. Simultaneously, persistent telomere damage activates chronic DNA-damage signaling that amplifies mitochondrial impairment and drives the accumulation of senescent cells. These senescent cells further perpetuate the cycle by releasing reactive oxygen species (ROS) and pro-inflammatory cytokines, thereby exacerbating oxidative injury, telomere attrition, and overall tissue aging.

To break this pathogenic feedback loop at its molecular origin, the study implemented an integrative therapeutic strategy combining Traditional Chinese Medicine (TCM) with targeted nutraceutical support. This dual approach was specifically designed to restore telomere stability, re-activate mitochondrial biogenesis, and mitigate cellular senescence through complementary mechanisms of action.

1. Traditional Chinese Medicine (TCM) Component

   Each participant received a sequential TCM regimen tailored to her reproductive profile and menstrual cycle phase:
   * Formula A ("Cycle Regulation & Pathogen Clearance") or "Endometrial Recovery & Mitochondrial Support", composed of Dan Shen, Dang Gui, Yu Jin, Hong Hua, and Ze Lan, was administered for 3-4 weeks to clear inflammatory stasis, enhance uterine microcirculation, and stimulate mitochondrial biogenesis through upregulation of PGC-1α and related transcriptional coactivators.
   * Formula B, administered in the luteal or preconception phase, focused on Kidney Yin-Yang repletion and endometrial priming, integrating Shu Di Huang, Tu Si Zi, Xu Duan, and Chuan Xiong to nourish oocytes, promote telomere stability, and support endocrine balance.

   Pharmacological studies have demonstrated that these botanical compounds modulate oxidative-stress pathways, telomerase activity, inflammatory mediators, and mitochondrial renewal, aligning with the biological mechanisms observed in "idiopathically" infertile women.
2. Nutraceutical Component

   In parallel, participants followed a nutraceutical protocol providing cofactors essential for telomere maintenance and mitochondrial energy metabolism, including Mito-PQQ, L-carnitine, Ubiquinol, Ω-3 PUFA, Resveratrol, N-acetyl-cysteine, Vitamin D3, B12, Zinc, and Magnesium. These molecules support ATP synthesis, redox homeostasis, DNA repair, and telomere stabilization, acting synergistically with the herbal formulations to reinforce cellular resilience.
3. Mechanistic Integration

Together, the TCM and nutraceutical interventions target multiple nodes of the aging network:

Telomere preservation, by reducing oxidative DNA damage and maintaining telomerase equilibrium;

Mitochondrial restoration, by reactivating biogenesis and improving energy metabolism;

Senescence reduction, by lowering oxidative stress, inflammatory signaling, and DNA-damage persistence.

This comprehensive approach aims to reverse the molecular hallmarks of reproductive aging, re-establishing cellular homeostasis and functional fertility potential in women previously classified as treatment-resistant.

6. Study Design and Objectives

This interventional clinical trial enrolled women aged 25-42 years with functionally idiopathic infertility, defined as post-treatment unexplained infertility following repeated failure of assisted reproductive technologies (ART) and other conventional interventions, despite adequate correction of known reproductive conditions. These women represent a clinically significant subgroup for whom infertility remains unexplained at the functional level but can now be biologically characterized through telomere-defined molecular aging profiles.

Study Phases

Baseline Assessment: Comprehensive reproductive evaluation and single-cell telomere profiling using the BEYOND GENOMiX FISH protocol to establish individual molecular signatures.

Pre-Conception Phase:

A 4- to 12-week personalized integrative protocol combining Traditional Chinese Medicine (TCM) herbal formulations with telomitochondrial-support nutraceuticals, tailored to each participant's telomere profile and menstrual phase.

Conception Attempt: Natural conception or ART (IUI/IVF) cycles conducted under continued integrative therapy to maintain telomere stability, enhance mitochondrial biogenesis, and reduce senescence-associated molecular stress.

Primary Objective

To evaluate whether telomere-guided integrative TCM therapy improves clinical pregnancy rates in women exhibiting telomere-defined molecular aging profiles after post-treatment ART failure.

Secondary Objectives

* To assess changes in telomere biomarkers (mean length, fraction of super-short telomeres, and overall distribution) after therapy.
* To evaluate ovarian reserve parameters (AMH, FSH, AFC), endometrial and menstrual characteristics, and overall safety and tolerability.
* To correlate molecular rejuvenation indicators (telomere restoration, mitochondrial function, and reduction in senescence) with reproductive outcomes, including fertilization, implantation, and sustained pregnancy.

This study design establishes a dynamic framework linking molecular aging biomarkers with reproductive outcomes, testing whether restoration of telomere integrity and its associated hallmarks of aging can translate into measurable fertility improvement in women with functionally idiopathic, post-treatment unexplained infertility.

ELIGIBILITY:
Inclusion Criteria:

* Biological female participants aged 25 to 42 years.
* Diagnosis of infertility defined as failure to conceive after at least 12 months of unprotected intercourse and/or repeated failure of assisted reproductive technologies (ART), including intrauterine insemination (IUI) and/or in vitro fertilization (IVF).
* History of post-treatment unexplained or functionally idiopathic infertility, defined as persistent infertility despite adequate correction or management of identifiable reproductive conditions (e.g., endometriosis, polycystic ovary syndrome, hormonal imbalance, uterine factors).
* Eligibility for natural conception attempts and/or assisted reproductive technologies according to routine clinical practice.
* Willingness to undergo biological aging biomarker profiling, including leukocyte telomere analysis.
* Ability and willingness to comply with study procedures, including the preconception integrative intervention and follow-up assessments.
* Provision of written informed consent prior to participation.

Exclusion Criteria:

* Current pregnancy or breastfeeding at the time of enrollment.
* Known chromosomal abnormalities or genetic conditions directly impairing fertility (e.g., Turner syndrome).
* Untreated severe male factor infertility precluding conception by natural or standard ART methods.
* Active malignancy or history of cancer requiring systemic treatment within the past 5 years.
* Severe systemic disease or medical condition contraindicating pregnancy or participation in ART (as determined by the treating physician).
* Use of investigational drugs or participation in another interventional clinical trial that could interfere with the study outcomes.
* Known hypersensitivity or contraindication to components of the integrative intervention, as determined by clinical assessment.
* Any condition which, in the opinion of the investigator, would interfere with safe participation or interpretation of study results.

Ages: 25 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate per Conception Attempt | From initiation of the conception attempt until confirmation of clinical pregnancy, assessed up to 12 months.
  Clinical pregnancy defined as the presence of an intrauterine gestational sac confirmed by transvaginal ultrasound following a natural conception attempt or assisted reproductive technology (IUI or IVF) cycle.

SECONDARY OUTCOMES:
Change in Percentage of Critically Short Telomeres (<5 kb) | Assessed from baseline to 3 months after initiation of the integrative intervention; participants without sufficient biological response at 3 months may undergo a second assessment at 6 months.
  Change from baseline in the percentage of leukocytes carrying critically short (super-short) telomeres shorter than 5 kilobases.
Change in Telomere Length Distribution Profile | Assessed from baseline to 3 months after initiation of the integrative intervention; participants without sufficient biological response at 3 months may undergo a second assessment at 6 months.
  Change from baseline in telomere length distribution patterns across individual leukocytes, assessed by single-cell FISH, including shifts toward shorter or longer telomere populations.
Change in Mean Leukocyte Telomere Length | From baseline to 3 months after initiation of the integrative intervention, with an additional assessment at 6 months if the biological response at 3 months is insufficient.
  Change from baseline in mean telomere length measured in peripheral blood leukocytes using single-cell FISH analysis.
Change in Serum Anti-Müllerian Hormone (AMH) Level | From baseline to 3 months after initiation of the integrative intervention, with an additional assessment at 6 months if the biological response at 3 months is insufficient.
  Change from baseline in serum AMH concentration, measured in ng/mL.
Change in Serum Follicle-Stimulating Hormone (FSH) Level | From baseline to 3 months after initiation of the integrative intervention, with an additional assessment at 6 months if the biological response at 3 months is insufficient.
  Change from baseline in serum FSH concentration, measured in IU/L.
Change in Antral Follicle Count (AFC) | Assessed from baseline to 3 months after initiation of the integrative intervention; participants without sufficient biological response at 3 months may undergo a second assessment at 6 months.
  Change from baseline in antral follicle count, reported as the number of antral follicles observed by transvaginal ultrasound.
Safety and Tolerability of the Integrative Intervention | From initiation of the integrative intervention through study completion (up to 12 months).
  Incidence of adverse events, abnormal laboratory findings, and treatment discontinuations related to the integrative intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- BEYOND GENOMiX Research and Coordination Center, Neuchâtel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bowen HJ. The determination of tin in biological material by using neutron-activation analysis. Analyst. 1972 Dec;97(161):1003-5. doi: 10.1039/an9729701003. No abstract available. PMID 4651952
- [Background] Ozturk S. The close relationship between oocyte aging and telomere shortening, and possible interventions for telomere protection. Mech Ageing Dev. 2024 Apr;218:111913. doi: 10.1016/j.mad.2024.111913. Epub 2024 Feb 1. PMID 38307343
- [Background] Zhou X, Smith DL, Lin J, HogenEsch E, Cedars MI. Telomere Length, Psychological Stress, and Infertility in Women of Advanced Reproductive Age. Endocrinology. 2025 Nov 6;166(12):bqaf163. doi: 10.1210/endocr/bqaf163. PMID 41233938
- [Background] Ruth KS, Day FR, Hussain J, Martinez-Marchal A, Aiken CE, Azad A, Thompson DJ, Knoblochova L, Abe H, Tarry-Adkins JL, Gonzalez JM, Fontanillas P, Claringbould A, Bakker OB, Sulem P, Walters RG, Terao C, Turon S, Horikoshi M, Lin K, Onland-Moret NC, Sankar A, Hertz EPT, Timshel PN, Shukla V, Borup R, Olsen KW, Aguilera P, Ferrer-Roda M, Huang Y, Stankovic S, Timmers PRHJ, Ahearn TU, Alizadeh BZ, Naderi E, Andrulis IL, Arnold AM, Aronson KJ, Augustinsson A, Bandinelli S, Barbieri CM, Beaumont RN, Becher H, Beckmann MW, Benonisdottir S, Bergmann S, Bochud M, Boerwinkle E, Bojesen SE, Bolla MK, Boomsma DI, Bowker N, Brody JA, Broer L, Buring JE, Campbell A, Campbell H, Castelao JE, Catamo E, Chanock SJ, Chenevix-Trench G, Ciullo M, Corre T, Couch FJ, Cox A, Crisponi L, Cross SS, Cucca F, Czene K, Smith GD, de Geus EJCN, de Mutsert R, De Vivo I, Demerath EW, Dennis J, Dunning AM, Dwek M, Eriksson M, Esko T, Fasching PA, Faul JD, Ferrucci L, Franceschini N, Frayling TM, Gago-Dominguez M, Mezzavilla M, Garcia-Closas M, Gieger C, Giles GG, Grallert H, Gudbjartsson DF, Gudnason V, Guenel P, Haiman CA, Hakansson N, Hall P, Hayward C, He C, He W, Heiss G, Hoffding MK, Hopper JL, Hottenga JJ, Hu F, Hunter D, Ikram MA, Jackson RD, Joaquim MDR, John EM, Joshi PK, Karasik D, Kardia SLR, Kartsonaki C, Karlsson R, Kitahara CM, Kolcic I, Kooperberg C, Kraft P, Kurian AW, Kutalik Z, La Bianca M, LaChance G, Langenberg C, Launer LJ, Laven JSE, Lawlor DA, Le Marchand L, Li J, Lindblom A, Lindstrom S, Lindstrom T, Linet M, Liu Y, Liu S, Luan J, Magi R, Magnusson PKE, Mangino M, Mannermaa A, Marco B, Marten J, Martin NG, Mbarek H, McKnight B, Medland SE, Meisinger C, Meitinger T, Menni C, Metspalu A, Milani L, Milne RL, Montgomery GW, Mook-Kanamori DO, Mulas A, Mulligan AM, Murray A, Nalls MA, Newman A, Noordam R, Nutile T, Nyholt DR, Olshan AF, Olsson H, Painter JN, Patel AV, Pedersen NL, Perjakova N, Peters A, Peters U, Pharoah PDP, Polasek O, Porcu E, Psaty BM, Rahman I, Rennert G, Rennert HS, Ridker PM, Ring SM, Robino A, Rose LM, Rosendaal FR, Rossouw J, Rudan I, Rueedi R, Ruggiero D, Sala CF, Saloustros E, Sandler DP, Sanna S, Sawyer EJ, Sarnowski C, Schlessinger D, Schmidt MK, Schoemaker MJ, Schraut KE, Scott C, Shekari S, Shrikhande A, Smith AV, Smith BH, Smith JA, Sorice R, Southey MC, Spector TD, Spinelli JJ, Stampfer M, Stockl D, van Meurs JBJ, Strauch K, Styrkarsdottir U, Swerdlow AJ, Tanaka T, Teras LR, Teumer A, Thornorsteinsdottir U, Timpson NJ, Toniolo D, Traglia M, Troester MA, Truong T, Tyrrell J, Uitterlinden AG, Ulivi S, Vachon CM, Vitart V, Volker U, Vollenweider P, Volzke H, Wang Q, Wareham NJ, Weinberg CR, Weir DR, Wilcox AN, van Dijk KW, Willemsen G, Wilson JF, Wolffenbuttel BHR, Wolk A, Wood AR, Zhao W, Zygmunt M; Biobank-based Integrative Omics Study (BIOS) Consortium; eQTLGen Consortium; Biobank Japan Project; China Kadoorie Biobank Collaborative Group; kConFab Investigators; LifeLines Cohort Study; InterAct consortium; 23andMe Research Team; Chen Z, Li L, Franke L, Burgess S, Deelen P, Pers TH, Grondahl ML, Andersen CY, Pujol A, Lopez-Contreras AJ, Daniel JA, Stefansson K, Chang-Claude J, van der Schouw YT, Lunetta KL, Chasman DI, Easton DF, Visser JA, Ozanne SE, Namekawa SH, Solc P, Murabito JM, Ong KK, Hoffmann ER, Murray A, Roig I, Perry JRB. Genetic insights into biological mechanisms governing human ovarian ageing. Nature. 2021 Aug;596(7872):393-397. doi: 10.1038/s41586-021-03779-7. Epub 2021 Aug 4. PMID 34349265
- [Background] M'kacher R, Colicchio B, Marquet V, Borie C, Najar W, Hempel WM, Heidingsfelder L, Oudrhiri N, Al Jawhari M, Wilhelm-Murer N, Miguet M, Dieterlen A, Deschenes G, Tabet AC, Junker S, Grynberg M, Fenech M, Bennaceur-Griscelli A, Voisin P, Carde P, Jeandidier E, Yardin C. Telomere aberrations, including telomere loss, doublets, and extreme shortening, are increased in patients with infertility. Fertil Steril. 2021 Jan;115(1):164-173. doi: 10.1016/j.fertnstert.2020.07.005. Epub 2020 Dec 4. PMID 33272625
- [Background] Lopez-Otin C, Blasco MA, Partridge L, Serrano M, Kroemer G. The hallmarks of aging. Cell. 2013 Jun 6;153(6):1194-217. doi: 10.1016/j.cell.2013.05.039. PMID 23746838